CLINICAL TRIAL: NCT05179759
Title: Teacher-delivered Transdiagnostic Child Mental Healthcare in Rural Primary Schools in India: a Batched Stepped-wedge Cluster Randomized Controlled Trial With a Hybrid Effectiveness-implementation-context Design
Brief Title: Teachers Leading the Frontlines (Tealeaf) - a Hybrid Effectiveness, Implement, and Context Trial
Acronym: Tealeaf
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Mariwala Health Initiative (Unknown); Colorado School of Public Health (Other); University of North Bengal (Unknown); University of Houston (Other); Broadleaf Health and Education Alliance (Other); Darjeeling Ladenla Road Prerna (DLRP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-2499; CTRI/2022/02/040398 (Registry Identifier: CTR-I (Clinical Trials Registry-India))
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Child Behavior Disorders
Keywords: child; child behavior; child behavior disorders; global health; India; mental health; schools; school mental health services; school teachers/psychology; students/psychology; child mental health; school-based intervention; task shifting; teacher-delivered care; stepped-wedge cluster randomized trial; implementation science; transdiagnostic intervention; mixed-methods research; rural health
MeSH Terms: conditions — Child Behavior Disorders; Child Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a batched stepped-wedge cluster randomized trial. Given the nature of the intervention, each school will be a cluster and each step will be an academic year. Schools will be enrolled into one of two batches and randomization will occur at the school level with multiple sequences within each batch. All schools will initially receive the control condition (EUC) and will be randomly and sequentially transitioned into the intervention arm. A qualitative exploration of context and process will be embedded within the framework of the randomized control trial, consistent with a hybrid effectiveness-implementation-context design. An embedded approach has been chosen to facilitate a high level of integration between the qualitative and quantitative components of the study.
Who Masked: Outcomes Assessor
Masking Description: Complete double-blinding is not possible in this cluster randomized stepped-wedge mental health intervention trial as trial participants and the intervention team will be aware of their status (open-label at the school and teacher level). However, to minimize bias and the risk of unmasking, the field team will be separated into intervention and data collection teams. The data collection team will be blinded to intervention allocation at the cluster-level and to treatment status at the individual child level. Additionally, while over time it may be likely that children and caregivers are aware of the intervention delivered, they will not be explicitly informed of this allocation. Outcome assessors will remain blinded throughout data collection. The study statistician will be unblinded for analysis purposes but will have no contact with study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Tealeaf - Year 1: Clusters (schools) and associated participants assigned to EUC (control) (Active Comparator): Clusters (schools) and associated participants are all assigned to the EUC condition in the 1st year of trial participation and transition to Tealeaf condition in subsequent years based on randomization assignment to 1 of 6 sequences in 1 of 2 batches.
  Interventions: Behavioral: Enhanced Usual Care
- Tealeaf - Year 1: Clusters (schools) and associated participants assigned to Tealeaf (experimental) (Experimental): Active intervention: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family. In Year 1, no schools are assigned to Tealeaf; schools transition to Tealeaf in subsequent years based on randomized assignment to 1 of 6 sequences and 1 of 2 batches.
  Interventions: Behavioral: Tealeaf
- Tealeaf - Year 2: Clusters (schools) and associated participants assigned to EUC (control) (Active Comparator): Enhanced Usual Care (EUC) is a less intensive version of the Tealeaf intervention. The EUC service package has been designed to be the most intensive form of care that could be envisioned as viable in the study setting in the foreseeable future without a significant increase in resource investment. Based on randomization assignment, clusters (schools) and associated participants that are in the active comparator arm receive EUC condition in Year 2 of the trial.
  Interventions: Behavioral: Enhanced Usual Care
- Tealeaf - Year 2: Clusters (schools) and associated participants assigned to Tealeaf (experimental) (Experimental): Active intervention: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family. In Year 2, based on randomization assignment, clusters (schools) and associated participants that are in the experimental arm receive Tealeaf intervention.
  Interventions: Behavioral: Tealeaf
- Tealeaf - Year 3: Clusters (schools) and associated participants assigned to EUC (control) (Active Comparator): Enhanced Usual Care (EUC) is a less intensive version of the Tealeaf intervention. The EUC service package has been designed to be the most intensive form of care that could be envisioned as viable in the study setting in the foreseeable future without a significant increase in resource investment. Based on randomization assignment, clusters (schools) and associated participants that are in the active comparator arm receive EUC condition in Year 3 of the trial.
  Interventions: Behavioral: Enhanced Usual Care
- Tealeaf - Year 3: Clusters (schools) and associated participants assigned to Tealeaf (experimental) (Experimental): Active intervention: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family. In Year 3, based on randomization assignment, clusters (schools) and associated participants that are in the experimental arm receive Tealeaf intervention.
  Interventions: Behavioral: Tealeaf
- Tealeaf - Year 4: Clusters (schools) and associated participants assigned to EUC (control) (Active Comparator): Enhanced Usual Care (EUC) is a less intensive version of the Tealeaf intervention. The EUC service package has been designed to be the most intensive form of care that could be envisioned as viable in the study setting in the foreseeable future without a significant increase in resource investment. Based on randomization assignment, clusters (schools) and associated participants that are in the active comparator arm receive EUC condition in Year 4 of the trial.
  Interventions: Behavioral: Enhanced Usual Care
- Tealeaf - Year 4: Clusters (schools) and associated participants assigned to Tealeaf (experimental) (Experimental): Active intervention: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family. In Year 4, based on randomization assignment, clusters (schools) and associated participants that are in the experimental arm receive Tealeaf intervention.
  Interventions: Behavioral: Tealeaf
- Tealeaf - Year 5: Clusters (schools) and associated participants assigned to EUC (control) (Active Comparator): Enhanced Usual Care (EUC) is a less intensive version of the Tealeaf intervention. The EUC service package has been designed to be the most intensive form of care that could be envisioned as viable in the study setting in the foreseeable future without a significant increase in resource investment. In Year 5, all schools have transitioned to Tealeaf. No schools are in the comparator arm.
  Interventions: Behavioral: Enhanced Usual Care
- Tealeaf - Year 5: Clusters (schools) and associated participants assigned to Tealeaf (experimental) (Experimental): Active intervention: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family. In Year 5, all clusters (schools) and associated participants are in the experimental arm and receive Tealeaf intervention.
  Interventions: Behavioral: Tealeaf

INTERVENTIONS:
Behavioral: Tealeaf — Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family.
  Arms: Tealeaf - Year 1: Clusters (schools) and associated participants assigned to Tealeaf (experimental); Tealeaf - Year 2: Clusters (schools) and associated participants assigned to Tealeaf (experimental); Tealeaf - Year 3: Clusters (schools) and associated participants assigned to Tealeaf (experimental); Tealeaf - Year 4: Clusters (schools) and associated participants assigned to Tealeaf (experimental); Tealeaf - Year 5: Clusters (schools) and associated participants assigned to Tealeaf (experimental)
Behavioral: Enhanced Usual Care — Enhanced Usual Care (EUC) is a less intensive version of the Tealeaf intervention. The EUC service package has been designed to be the most intensive form of care that could be envisioned as viable in the study setting in the foreseeable future without a significant increase in resource investment
  Other Names: EUC
  Arms: Tealeaf - Year 1: Clusters (schools) and associated participants assigned to EUC (control); Tealeaf - Year 2: Clusters (schools) and associated participants assigned to EUC (control); Tealeaf - Year 3: Clusters (schools) and associated participants assigned to EUC (control); Tealeaf - Year 4: Clusters (schools) and associated participants assigned to EUC (control); Tealeaf - Year 5: Clusters (schools) and associated participants assigned to EUC (control)

SUMMARY:
Purpose: The overall aim of this study is to evaluate the effectiveness, implementation, and contextual influences of a teacher-delivered transdiagnostic model of child mental health care (Tealeaf) for school-aged children in resource-limited primary schools in the Darjeeling Himalayas.

Participants: Within 90 rural, low-cost private primary schools across the Darjeeling and Kalimpong districts of the Indian Himalayas, all teachers meeting eligibility criteria will be invited to participate in training and the intervention. The number of teachers consented and enrolled into the study will be determined by the size of the school. The number of students nominated by a teacher is at their discretion (including an option to not nominate any student in a given year if they do not perceive any of the students to be appropriate for the intervention) However, based on the research team's pilot data and prior experience, teachers will be provided with the suggestion that they nominate two children to receive targeted intervention. For each child receiving intervention, a paired parent or guardian will be recruited and enrolled to the study.

Procedures (methods): Effectiveness will be evaluated through a botched stepped-wedge cluster randomized controlled trial with an embedded mixed methods evaluation of implementation and qualitative study of context (guided by the RE-AIM framework). Schools will begin in enhanced usual care (EUC) and cross over to the Tealeaf intervention as per a randomized schedule. In Batch 1, year 1 will include 60 schools in the control arm, year 2 will include 40 schools in the control arm and 20 in the intervention arm, year 3 will include 20 schools in the control arm and 40 in the intervention arm, and year 4 will include 60 schools in the intervention arm. Batch 2 will be operationalized in the third year of the study. In Batch 2, year 3 will include 30 schools in the control arm, year 4 will include 10 schools in the control arm and 20 schools in the intervention arm, and year 5 will include 30 schools in the intervention arm. The primary effectiveness outcome is teacher-reported child mental health status; secondary outcomes include parent-reported symptoms, adaptive functioning, academic achievement, and attendance. Implementation outcomes will be assessed using the RE-AIM framework. A parallel qualitative study will generate contextual understanding through longitudinal ethnography, interviews, participant observation, and field notes.

DETAILED DESCRIPTION:
Expanding access to children's mental health care is a critically important global health challenge. Twenty percent of all children suffer from significant mental health concerns, most of whom will remain unrecognized, unsupported and affected throughout their lives. In India and low and middle income countries (LMICs), the burden of children's mental illness is particularly heavy due to large populations with high proportions of children and adolescents, high rates of adverse childhood events and poverty, limited resources to care for children and under-recognition of their mental health struggles. Despite prevalence rates in India estimated to be on the high end of the global burden, less than 1% of Indian children and adolescents with mental health struggles are receiving treatment. The need to address this care gap is further intensified by the adverse impacts of the Covid-19 pandemic. Task-shifting of mental health care tasks to non-specialist providers and lay individuals in LMICs has been shown repeatedly to increase access to care and improve mental health outcomes; it represents a promising approach to delivery of child mental healthcare. However, alternative models for children's mental healthcare, including task-shifting, are rare and reflect several significant barriers. Provision of such care occurring in the context of children's evolving cognitive and emotion-recognition abilities requires knowledge of and experience in child development. Furthermore, given limited funding and few professional providers for children's mental health, sustainable care models likely need to leverage existing systems and require few or no additional human resources. With relevant professional experience and consistent access to children within existing education systems, teachers are uniquely positioned to address these barriers and deliver care to children. School-based mental health interventions are commonly conceptualized using the Multi-Tiered Systems of Support (MTSS) framework which defines three levels of support corresponding with Tier 1(promotion), Tier 2 (prevention), and Tier 3 (intervention & treatment). Several studies have demonstrated that teachers can successfully deliver whole-school or whole-class-based interventions targeting universal mental health prevention and promotion in resource-constrained settings. Far fewer efforts, however, have been undertaken to evaluate the possibility of Tier 3 interventions in which teachers directly provide care to select children-in-need. Teachers in an HIC have been able to feasibly deliver a subset of therapeutic techniques to children diagnosed with Conduct Disorder and an ongoing study in Kenya has shown teacher-delivered Trauma-focused-Cognitive Behavioral Therapy for children who have experienced parental death is feasible and acceptable. While these studies suggest promise for teacher-delivered indicated care, teachers in these handful of studies delivered prescribed, manualized care. While such a structure is at the heart of task-shifted care for adults and adolescents, it differs from the typical Tier 1 and Tier 2 structure that is either whole-school or whole-class-based. It may be that few interventions study teachers delivering Tier 3 care as the typical Tier 3 structure, predominantly one-on-one sessions, is not conducive to teachers delivering care on top of their typical duties. Further, the care in these studies focuses on singular diagnoses, limiting the teacher-lay counselors' reach. Given the limited time teacher-lay counselors would have to deliver indicated care, a transdiagnostic approach would maximize the children and categories of struggles teachers could reach while potentially minimizing the amount of training teachers would need to deliver such care. To address this gap, the research team has developed a novel intervention, Tealeaf, to task-shift to to teachers the delivery of care to indicated school-aged children facing mental distress. Tealeaf is unique in that teachers deliver care utilizing a trans-diagnostic, non-manualized, evidence-based approach that they can customize and integrate into their existing workflows. In work preceding this trial, members of this research group conducted studies in rural Darjeeling to assess the feasibility, acceptability and potential efficacy of Tealeaf. Through this work, the research team has documented an emergent therapy modality that they have called "education as mental health therapy" (Ed-MH). Ed-MH relies on teachers shifting their professional practice to incorporate mental health techniques into their workflow with the primary goal of improving individual children's mental wellbeing. Transdiagnostic, indicated mental health care that is primarily incorporated into existing workflows is feasible for teachers to deliver and acceptable to teachers, caregivers, and children. Further, the research team has established strong face validity for the efficacy of Tealeaf. Children receiving this care have consistently demonstrated significant improvement in their mental health from baseline and an (ad-hoc) showed substantial/significant impact for children receiving Tealeaf as compared to Enhanced Usual Care [publication forthcoming]. Finally, the potential risks associated with Tealeaf have been well evaluated and no serious adverse events have occurred over multiple years of piloting. Overall, the research team's prior research demonstrates that teacher-delivered transdiagnostic mental health care (Ed-MH) may be a potentially efficient, sustainable, and impactful approach. The research team believes the next logical step is to assess the effectiveness of this care model through real-world implementation. To accomplish this, with funding support from the Mariwala Health Initiative, the research team will conduct a hybrid three-variable hybrid study of effectiveness, implementation, and context. Evaluating intervention effectiveness, implementation processes and outcomes, and the context in which it occurs will generate valuable insight into how children's mental health care can best be delivered in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

Clusters (schools):

* Does not receive government aid (i.e., not subject to the rules and regulations of government or government-aided schools,
* At least 3 full-time classroom teachers on staff,
* Annual student fees $200/14,500 Indian rupee (INR) or less
* Low-cost private primary schools in rural Darjeeling and Kalimpong districts

Teachers:

* Employed at a participating school,
* Have primary teaching responsibility in the primary grade level,
* Are 18 years or older

Children:

* Enrolled in class I-IV,
* Enrolled in the classroom of a participating teacher

Exclusion Criteria:

Clusters (schools):

* Not located in urban areas of the Darjeeling and Kalimpong Districts defined as the statutory towns of Darjeeling, Kurseon, Mirik and the Kalimpong Municipality.

Teachers:

* Have been convicted and/or are under investigation for any child-related misconduct or maltreatment.

Children:

* Do not have a parent or guardian who can provide informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20160 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean Difference on the Achenbach System of Empirically Based Assessment (ASEBA) Teacher Report Form Total Problem Scale | 8 months from baseline
  The ASEBA TRF is a standardized tool to assess school adaptive function in children. Teachers rate the child on 7-point scales in four areas: how hard he/she is working, how appropriately he/she is behaving, how much he/she is learning, and how happy he/she is. Raw and T-scores on the Adaptive Functioning Scale are derived from the sum of the individual items. A higher score indicates better school adaptive function.

SECONDARY OUTCOMES:
Mean Difference at Endline on the Strengths and Difficulties Questionnaire Total Difficulties Score | 8 months from baseline
  The Strengths and Difficulties Questionnaire Total is a standardized tool to measure for psychopathology in children and adolescents. A Total Difficulties scale score is derived by summing items from four problem subscales (emotional, conduct, hyperactivity/inattention, and peer relationship), while a fifth subscale (prosocial functioning) does not contribute to the overall severity score. Scores also include an internalizing score, externalizing score, and impact score. Individual problem scale items are scored from 0 to 2 (with higher scores indicating greater problem severity).
Mean Difference on Annual Status of Education Report (ASER) Composite Score | 8 months from baseline
  The ASER is a measure of academic performance of children 6-14 in India. Domains assessed include reading, math, and English. The tool was expanded to include assessment of higher-order functions. A composite score is derived from the score on individual assessment domains. The ranges for each domain are as follows: Math (0-10), Reading (0-5), Total (0-15). A higher score indicated that the child scored at a higher grade level.
Mean Difference in Proportion of School Days Absent | 8 months from baseline
  School attendance data will be obtained from teacher-completed and school-maintained log books of student attendance. Given that the school year varies by school, the number of days a child is absent will be converted to a proportion.
TRF Adaptive Functioning | 8 months from baseline
  The ASEBA Teacher Report Form (TRF) uses standardized norms to measure child functioning with high reliability and validity. The TRF adaptive functioning instrument documents children's scores on a 7-point response scale: work effort, behavioral appropriateness, learning, and happiness. Teachers rate each item on a 7-point scale. Scores from the four subscales are summed, and T-scores are used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Cruz, MD, EdM, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- DLR Prerna, Darjeeling, West Bengal, India

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) generated during and/or analyzed during the study will not be publicly available including in de-identified form due to the potential for deductive disclosure, but may be available on reasonable request, subject to approval by Darjeeling Ladenla Road Prerna (DLRP) and DLRP governance.